CLINICAL TRIAL: NCT00386074
Title: The Efficacy of Iron Fortified Whole Maize Flour on the Iron Status of School Children in Kenya
Brief Title: Iron-fortified Whole Maize Flour Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Unilever Food and Health Research Institute, The Netherlands (Unknown); Kenya Medical Research Institute (Other); Akzo Nobel (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6107050200
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2010-04-21 (Estimated); Status verified 2010-04

CONDITIONS: Anaemia
Keywords: NaFeEDTA; electrolytic iron; efficacy; whole maize flour; phytate; school-age children; controlled trial; Africa
MeSH Terms: conditions — Anemia | interventions — Fe(III)-EDTA

INTERVENTIONS:
Drug: NaFeEDTA, Electrolytic Iron

SUMMARY:
The purpose of this study is to assess whether NaFeEDTA and electrolytic iron improve iron status of young school children, when added as iron fortificants in whole maize flour.

DETAILED DESCRIPTION:
Fortification of staple foods with iron may be an effective method of addressing the problem of iron deficiency. Questions however remain of the type of iron fortificants to use, the appropriate fortification levels and suitable food vehicles. Cereals form attractive vehicles because they are widely consumed in parts of the world that bear a large burden of the iron deficiency problem. They are however high in phytates and would reduce the bioavailability of commonly used iron fortificants. Isotope studies have shown that even in the presence of phytates, iron from NaFeEDTA is relatively more bioavailable than that from other fortificant sources. Its efficacy has however not been assessed in human trials. Electrolytic iron, on the other hand is widely used and was legislated as the iron fortificant of choice in South Africa. Its efficacy in a high-phytate vehicle has also not been assessed. We have therefore undertaken to assess the efficacy of NaFeEDTA at two doses, as an iron fortificant in whole flour, and the efficacy of electrolytic iron at a dose similar to the high-dose NaFeEDTA. The results will contribute information on the suitability of these fortificants in whole maize flour, a food commonly consumed in sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:Children:

* 3-8 years age (for the purposes of this study this will include children born within the period December 15th 1995- May 1st 2001).
* Whohave been resident in the area for 6 months or more.
* Enrolled in the selected schools
* Able to consume the target amount of porridge, at least 50% of the time during the run-in period
* Will be present in the study area for the entire study period (April - December 2004).

Exclusion Criteria:

* Children below 3 years and above 8 years of age (born after December 15th 1995 and before May 1st 2001).
* Children who have been resident in the area for less than 6 months at the time of recruitment.
* Children with obvious physical and mental disability.
* Severely malnourished children.
* Severely anaemic children (Hb <70g/L).

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 412
Dates: Start 2004-05; Study Completion 2004-12

PRIMARY OUTCOMES:
Haemoglobin
Plasma Ferritin
Plasma Transferrin receptor

SECONDARY OUTCOMES:
Iron deficiency anaemia
Iron deficiency
Anaemia

CONTACTS AND LOCATIONS:
Overall Officials: Pauline EA Andang'o, MND, Principal Investigator — Wageningen University; David L Mwaniki, PhD, Principal Investigator — Kenya Medical Research Institute; Hans Verhoef, PhD, Principal Investigator — Wageningen University; Saskia JM Osendarp, PhD, Study Director — Unilever Food and Health Institute, Vlaardingen, The Netherlands; Frans J Kok, PhD, Study Chair — Wageningen University

REFERENCES:
- [Derived] Andang'o PE, Osendarp SJ, Ayah R, West CE, Mwaniki DL, De Wolf CA, Kraaijenhagen R, Kok FJ, Verhoef H. Efficacy of iron-fortified whole maize flour on iron status of schoolchildren in Kenya: a randomised controlled trial. Lancet. 2007 May 26;369(9575):1799-1806. doi: 10.1016/S0140-6736(07)60817-4. PMID 17531887